CLINICAL TRIAL: NCT01301313
Title: Phase II Study to Evaluate the Efficacy and Safety of Levosimendan in Severe Acute Heart Failure in Critical Children
Brief Title: Efficacy and Safety of Levosimendan in Severe Acute Heart Failure in Critical Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Jose Luis Vazquez Martinez (Other)
Responsible Party: Sponsor-Investigator, Jose Luis Vazquez Martinez, Doctor, Hospital Universitario Ramon y Cajal
Organization: Hospital Universitario Ramon y Cajal (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LEVOPED1; 2009-017827-24 (EudraCT Number)
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Acute Heart Failure
Keywords: Acute heart failure; Children; Levosimendan; Inotropic treatment
MeSH Terms: interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levosimendan (Experimental)
  Interventions: Drug: Levosimendan
- Conventional intensified inotropic treatment (Active Comparator)
  Interventions: Drug: Conventional intensified inotropic treatment

INTERVENTIONS:
Drug: Levosimendan — Levosimendan 2.5 mg / ml ampoules. The drug will be administrated in continuous intravenous perfusion in a single dose of 0.1 - 0.2 micrograms/ kg / min for 24 hours.
  Arms: Levosimendan
Drug: Conventional intensified inotropic treatment — Increasing the dose and / or the number of inotropes (dopamine and / or dobutamine and / or milrinone and / or adrenaline)
  Arms: Conventional intensified inotropic treatment

SUMMARY:
To evaluate the efficacy and safety of levosimendan versus conventional intensified inotropic treatment, in critical children with severe acute heart failure which persists despite of having received conventional inotropic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written consent to participate in the study and for the transfer of material for cellular and molecular studies.
* Understand the purpose of the study and to be available to perform the procedures written in the protocol.
* Any child of 1 day old to 18 years old, admitted to the Paediatric Intensive Care Unit due to severe acute heart failure of any etiology.

Exclusion Criteria:

All patients who

* express their wish of not to participate in the protocol
* have hypertrophic or restrictive cardiomyopathy
* have aortic Stenosis
* have a known allergy to any drug used in the study
* it is not possible to prescribe the study medication because it is contraindicated according to the Summary of the Product Characteristic or according to the criteria of the physician responsible for patient
* are pregnant

Ages: 24 Hours to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Hemodynamic improvement at 24 hours | 24 hours
  To evaluate the efficacy of levosimendan in the treatment of severe acute heart failure in children in critical conditions comparing the proportion of patients with hemodynamic improvement at 24 hours between the group who received levosimendan as rescue therapy (experimental treatment) versus the one who received intensified conventional inotropic treatment (control treatment)

SECONDARY OUTCOMES:
Improvement in cardiac output | 24 and 48 hours
  To compare the improvement in cardiac output induced by levosimendan in the treatment of severe acute heart failure in critical children versus the intensified conventional inotropic treatment, at 24 and 48h
Improvement in the neurohormonal profile | 24 and 48 hours
  To compare the improvement in the neurohormonal profile (assessed as a reduction of BNP) induced by levosimendan in the treatment of severe acute heart failure in critical children versus the intensified conventional inotropic treatment, at 24 and 48h.
Number of days of hospital stay in paediatric intensive care unit | 30 days
  To compare the number of days of hospital stay in paediatric intensive care unit and the number of days on mechanical ventilation, at 30 days.
Safety | 30 days
  To assess the safety of the use of levosimendan in the treatment of severe acute heart failure in children in critical conditions, at 30 days.
Survival | 30 days
  Survival, at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Vazquez MArtinez, MD, Principal Investigator — Hospital Universitario Ramón y Cajal. Madrid
Locations (19):
- Spain (19):
  - Hospital Clínico Universitario de Santiago de Compostela, A Coruña, A Coruña
  - Hospital Juan Canalejo, A Coruña, A Coruña
  - Hospital San Joan de Deu, Barcelona, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Infantil La Paz, Madrid, Madrid
  - Hospital Universitario Doce de Octubre, Madrid, Madrid
  - Hospital Universitario Carlos Haya, Málaga, Malaga
  - Hospital Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Clínico Universitario Son Dureta, Palma de Mallorca, Palma de Mallorca
  - Complejo Hospitalario Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Donosti, Donostia / San Sebastian, San Sebastian
  - Hospital Virgen de la Salud, Toledo, Toledo
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid
  - Hospital de Cruces, Vizcaya, Vizcaya
  - Hospital Miguel Servet, Zaragoza, Zaragoza